CLINICAL TRIAL: NCT02588508
Title: Effectiveness of Warm Packs, Perineal Massage and Hands Off During Labour in the Perineal Outcomes.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Jânio do Nascimento Alves, Master Student, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0335932
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Perineal Tear
Keywords: perineal tear; pain; pelvic floor; Labour
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Warm packs (Experimental): The warm packs are held in the mother's perineum during birth. The warm packs are changed as needed to maintain warmth.
  Interventions: Procedure: Warm packs
- Perineal massage (Experimental): The perineal massage will be gently held in the longitudinal direction of the muscle fibers, with movements of the thumb and forefinger, like "count coins".
  Interventions: Procedure: Perineal massage
- Hands off (No Intervention): Hands off group does not receive any perineal manipulation and they are only observed.

INTERVENTIONS:
Procedure: Warm packs — : The warm packs are held in the mother's perineum during birth. The warm packs are changed as needed to maintain warmth.
  Arms: Warm packs
Procedure: Perineal massage — The perineal massage will be gently held in the longitudinal direction of the muscle fibers, with movements of the thumb and forefinger, like "count coins".
  Arms: Perineal massage

SUMMARY:
This study evaluates the effectiveness of warm packs, perineal massage and hands off, during labour, in the perineal outcomes. The perineal outcomes are perineal tears, grade of perineal tears, need of suture, perineal edema, perineal pain, use of drugs for perineal pain, and satisfaction with the technique used.

DETAILED DESCRIPTION:
This study is a randomised controled trial.

ELIGIBILITY:
Inclusion Criteria:

* parturient in active phase of labour
* single fetus at term (37-42 weeks)
* bent cephalic fetal presentation
* parity less than four children

Exclusion Criteria:

* use any perineal preparation techniques during pregnancy
* clinical indication for caesarean section

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Need of suture | 30 minutes
  Number of participants with perineal tear after vaginal delivery requiring suture (evaluated as yes or no).

SECONDARY OUTCOMES:
Grade of perineal tear | 30 minutes
  Perineal tear ranked 1st, 2nd, 3rd and 4th degree
perineal edema | 1 hour
  Perineal edema is scored 0-4 (0 = no edema; 4 = edema invades the perineal body) .
Perineal pain | 24 hours
  self reported ´perineal pain intensity. Perineal pain is scored 0-10 (0 = no pain; 10 = pain as bad as can be).
Use of drugs for perineal pain | 24 hours
  Number of participants using drugs for perineal pain at the time of 24 hours after vaginal delivery (evaluated as yes or no).
Satisfaction with the technique used | 24 hours
  Satisfaction of the woman with the technique used for perineal care. Satisfaction is scored 0-4 (0 = very satisfied; 4 = very dissatisfied)
Perineal tear | 30 minutes
  Number of participants with perineal tear after vaginal delivery (evaluated as yes or no).

CONTACTS AND LOCATIONS:
Overall Officials: Caroline WS Ferreira, PHD, Study Director — Universidade Federal de Pernambuco
Locations (1):
- UFPernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Background] Aasheim V, Nilsen AB, Lukasse M, Reinar LM. Perineal techniques during the second stage of labour for reducing perineal trauma. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD006672. doi: 10.1002/14651858.CD006672.pub2. PMID 22161407
- [Background] Albers LL, Sedler KD, Bedrick EJ, Teaf D, Peralta P. Midwifery care measures in the second stage of labor and reduction of genital tract trauma at birth: a randomized trial. J Midwifery Womens Health. 2005 Sep-Oct;50(5):365-72. doi: 10.1016/j.jmwh.2005.05.012. PMID 16154062
- [Background] Albers LL, Sedler KD, Bedrick EJ, Teaf D, Peralta P. Factors related to genital tract trauma in normal spontaneous vaginal births. Birth. 2006 Jun;33(2):94-100. doi: 10.1111/j.0730-7659.2006.00085.x. PMID 16732773
- [Background] Albers LL, Borders N. Minimizing genital tract trauma and related pain following spontaneous vaginal birth. J Midwifery Womens Health. 2007 May-Jun;52(3):246-53. doi: 10.1016/j.jmwh.2006.12.008. PMID 17467591
- [Background] Althabe F, Belizan JM, Bergel E. Episiotomy rates in primiparous women in Latin America: hospital based descriptive study. BMJ. 2002 Apr 20;324(7343):945-6. doi: 10.1136/bmj.324.7343.945. No abstract available. PMID 11964339
- [Background] AMORIM, M. M. R. DE et al. Assistência humanizada ao parto no Instituto de Saúde Elpídio de Almeida (ISEA): resultados maternos. Revista Saúde & Ciência, v. v. I, n. n. 1, p. 80 - 7, 2010.
- [Background] AMORIM, M. M. R. DE; PORTO, A. M. F.; SOUZA, A. S. R. Assistência ao segundo e terceiro períodos do trabalho de parto baseada em evidências. Femina, v. 38, n. 11, p. 583-91, 2010.
- [Background] Beckmann MM, Garrett AJ. Antenatal perineal massage for reducing perineal trauma. Cochrane Database Syst Rev. 2006 Jan 25;(1):CD005123. doi: 10.1002/14651858.CD005123.pub2. PMID 16437520
- [Background] Carroli G, Belizan J. Episiotomy for vaginal birth. Cochrane Database Syst Rev. 2000;(2):CD000081. doi: 10.1002/14651858.CD000081. PMID 10796120
- [Background] COELHO, L. F. S. O treino de flexibilidade muscular e o aumento da amplitude de movimento: uma revisão crítica da literatura. Revista de Desporto e Saúde, v. 4, n. 3, p. 61-72, 2007.
- [Background] de Souza Caroci da Costa A, Gonzalez Riesco ML. A comparison of "hands off" versus "hands on" techniques for decreasing perineal lacerations during birth. J Midwifery Womens Health. 2006 Mar-Apr;51(2):106-11. doi: 10.1016/j.jmwh.2005.10.017. PMID 16504907
- [Background] Dahlen HG, Homer CS, Cooke M, Upton AM, Nunn R, Brodrick B. Perineal outcomes and maternal comfort related to the application of perineal warm packs in the second stage of labor: a randomized controlled trial. Birth. 2007 Dec;34(4):282-90. doi: 10.1111/j.1523-536X.2007.00186.x. PMID 18021143
- [Background] Dahlen HG, Homer CS, Cooke M, Upton AM, Nunn RA, Brodrick BS. 'Soothing the ring of fire': Australian women's and midwives' experiences of using perineal warm packs in the second stage of labour. Midwifery. 2009 Apr;25(2):e39-48. doi: 10.1016/j.midw.2007.08.002. Epub 2007 Nov 26. PMID 18031878
- [Background] Elharmeel SM, Chaudhary Y, Tan S, Scheermeyer E, Hanafy A, van Driel ML. Surgical repair of spontaneous perineal tears that occur during childbirth versus no intervention. Cochrane Database Syst Rev. 2011 Aug 10;2011(8):CD008534. doi: 10.1002/14651858.CD008534.pub2. PMID 21833968
- [Background] Dahlen HG. Perineal warm compress reduces risk of third- and fourth- degree tears and should be part of second stage care. Evid Based Nurs. 2012 Oct;15(4):103-4. doi: 10.1136/ebnurs-2012-100685. Epub 2012 Jun 12. No abstract available. PMID 22691406
- [Background] FELICE, T.; SANTANA, L. Recursos fisioterapêuticos (crioterapia e termoterapia) na espasticidade: revisão de literatura. Rev Neurocienc, v. 17, n. 1, p. 57-62, 2009.
- [Background] Flynn P, Franiek J, Janssen P, Hannah WJ, Klein MC. How can second-stage management prevent perineal trauma? Critical review. Can Fam Physician. 1997 Jan;43:73-84. PMID 9626426
- [Background] Geranmayeh M, Rezaei Habibabadi Z, Fallahkish B, Farahani MA, Khakbazan Z, Mehran A. Reducing perineal trauma through perineal massage with vaseline in second stage of labor. Arch Gynecol Obstet. 2012 Jan;285(1):77-81. doi: 10.1007/s00404-011-1919-5. Epub 2011 May 26. PMID 21614497
- [Background] Helewa ME. Episiotomy and severe perineal trauma. Of science and fiction. CMAJ. 1997 Mar 15;156(6):811-3. No abstract available. PMID 9084387
- [Background] Howard D, Davies PS, DeLancey JO, Small Y. Differences in perineal lacerations in black and white primiparas. Obstet Gynecol. 2000 Oct;96(4):622-4. doi: 10.1016/s0029-7844(00)00956-x. PMID 11004370
- [Background] Klein MC, Gauthier RJ, Robbins JM, Kaczorowski J, Jorgensen SH, Franco ED, Johnson B, Waghorn K, Gelfand MM, Guralnick MS, et al. Relationship of episiotomy to perineal trauma and morbidity, sexual dysfunction, and pelvic floor relaxation. Am J Obstet Gynecol. 1994 Sep;171(3):591-8. doi: 10.1016/0002-9378(94)90070-1. PMID 8092203
- [Background] Klein MC, Janssen PA, MacWilliam L, Kaczorowski J, Johnson B. Determinants of vaginal-perineal integrity and pelvic floor functioning in childbirth. Am J Obstet Gynecol. 1997 Feb;176(2):403-10. doi: 10.1016/s0002-9378(97)70506-4. PMID 9065189
- [Background] LEAL, N. V et al. Factors associated with perineal lacerations requiring suture in vaginal births without episiotomy. Obstetrics and gynecology, v. 123 Suppl , p. 63S-4S, maio 2014.
- [Background] Lundquist M, Olsson A, Nissen E, Norman M. Is it necessary to suture all lacerations after a vaginal delivery? Birth. 2000 Jun;27(2):79-85. doi: 10.1046/j.1523-536x.2000.00079.x. PMID 11251483
- [Background] Macarthur AJ, Macarthur C. Incidence, severity, and determinants of perineal pain after vaginal delivery: a prospective cohort study. Am J Obstet Gynecol. 2004 Oct;191(4):1199-204. doi: 10.1016/j.ajog.2004.02.064. PMID 15507941
- [Background] Messelink B, Benson T, Berghmans B, Bo K, Corcos J, Fowler C, Laycock J, Lim PH, van Lunsen R, a Nijeholt GL, Pemberton J, Wang A, Watier A, Van Kerrebroeck P. Standardization of terminology of pelvic floor muscle function and dysfunction: report from the pelvic floor clinical assessment group of the International Continence Society. Neurourol Urodyn. 2005;24(4):374-80. doi: 10.1002/nau.20144. No abstract available. PMID 15977259
- [Background] OMS. Integrated management of pregnancy and childbirth. Manejo de las complicaciones del embarazo e el parto: Guía para obstetrices y médicos. OMS ed. Ginebra: [s.n.]. p. 438
- [Background] Patel DA, Xu X, Thomason AD, Ransom SB, Ivy JS, DeLancey JO. Childbirth and pelvic floor dysfunction: an epidemiologic approach to the assessment of prevention opportunities at delivery. Am J Obstet Gynecol. 2006 Jul;195(1):23-8. doi: 10.1016/j.ajog.2006.01.042. Epub 2006 Mar 30. PMID 16579934
- [Background] PHILLIPS, C.; MONGA, A. Childbirth and the pelvic floor: "the gynaecological consequences."Reviews in Gynaecological Practice, v. 5, n. 1, p. 15-22, mar. 2005.
- [Background] Rathfisch G, Dikencik BK, Kizilkaya Beji N, Comert N, Tekirdag AI, Kadioglu A. Effects of perineal trauma on postpartum sexual function. J Adv Nurs. 2010 Dec;66(12):2640-9. doi: 10.1111/j.1365-2648.2010.05428.x. Epub 2010 Aug 23. PMID 20735499
- [Background] Renfrew MJ, Hannah W, Albers L, Floyd E. Practices that minimize trauma to the genital tract in childbirth: a systematic review of the literature. Birth. 1998 Sep;25(3):143-60. doi: 10.1111/j.1523-536x.1998.t01-2-.x. PMID 9767217
- [Background] Sanders J, Peters TJ, Campbell R. Techniques to reduce perineal pain during spontaneous vaginal delivery and perineal suturing: a UK survey of midwifery practice. Midwifery. 2005 Jun;21(2):154-60. doi: 10.1016/j.midw.2004.12.003. Epub 2005 Mar 27. PMID 15878430
- [Background] SANTOS, J. DE O. et al. Freqüência de traumas perineais nos partos vaginais. Esc Anna Nery Rev Enferm, v. 12, n. 4, p. 658-63, 2008.
- [Background] Scott JR. Episiotomy and vaginal trauma. Obstet Gynecol Clin North Am. 2005 Jun;32(2):307-21, x. doi: 10.1016/j.ogc.2004.12.001. PMID 15899363
- [Background] Stamp G, Kruzins G, Crowther C. Perineal massage in labour and prevention of perineal trauma: randomised controlled trial. BMJ. 2001 May 26;322(7297):1277-80. doi: 10.1136/bmj.322.7297.1277. PMID 11375230
- [Background] TORRES, I. M. Efetividade da crioterapia para o controle da dor perineal no pós-parto vaginal imediato: ensaio clínico randomizado. 2013. Dissertação (Mestrado em Saúde Materno-Infantil). Instituto de Medicina Integral Professor Fernando Figueira, Recife, 2013.
- [Background] ZANETTI, M. R. D. et al. Episiotomia : revendo conceitos. Femina, v. 37, n. 7, p. 5-9, 2009.